CLINICAL TRIAL: NCT03069378
Title: A Phase II Study of Talimogene Laherparepvec (T-VEC) Administered Concurrently With the Anti-PD1 Monoclonal Antibody Pembrolizumab in Patients With Metastatic and/or Locally Advanced Sarcoma
Brief Title: A Study of Talimogene Laherparepvec (T-VEC) in Combination With Pembrolizumab in Patients With Metastatic and/or Locally Advanced Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1534
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma; Epithelioid Sarcoma; Cutaneous Angiosarcoma
Keywords: Metastatic; Locally Advanced; Talimogene Laherparepvec (T-VEC); Pembrolizumab; 16-1534
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — talimogene laherparepvec; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a single-center, phase II study to evaluate the efficacy of the oncolytic herpes virus talimogene laherparepvec, given in combination with pembrolizumab for patients with metastatic and/or locally advanced sarcomas.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talimogene Laherparepvec (T-VEC) Administered with Pembrolizu (Experimental): Patients will initiate treatment with talimogene laherparepvec given intralesionally and pembrolizumab.
  Interventions: Drug: Talimogene Laherparepvec (T-VEC); Drug: Pembrolizumab

INTERVENTIONS:
Drug: Talimogene Laherparepvec (T-VEC) — Talimogene laherparepvec treatment will be given at Day 1 Week 1, and every 3 weeks thereafter .
Drug: Pembrolizumab — Pembrolizumab will be given at Day 1 week 1 and every 3 weeks thereafter.

SUMMARY:
The purpose of this study is to determine how well the combination of therapy of talimogene laherparepvec (T-VEC) and pembrolizumab works in the treatment of patients with sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years at the time of informed consent
* Be willing and able to provide written informed consent/assent for the trial
* Be willing to comply with treatment protocol
* Subjects must have a histologically confirmed metastatic and/or locally advanced inoperable sarcoma (metastatic/locally advanced cohort)
* For histology specific additional metastatic cohorts, patients must have undifferentiated pleomorphic sarcoma/myxofibrosarcoma, epithelioid sarcoma or cutaneous angiosarcoma.
* Subjects must have at least 1 injectable cutaneous, subcutaneous (superficial or deep) soft tissue or nodal lesion ≥ 10 mm in longest diameter. Of note, bone lesions are not eligible for injection unless there is a soft tissue component that is amenable to injection. Injectable lesions must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment
* Subjects with locally advanced/metastatic sarcoma must have at least one prior line of systemic therapy (e.g. chemotherapy, immunotherapy, targeted or biological therapy). An exception to this criterion will be made for patients with sarcoma histological subtypes for which there is no known standard systemic therapy (e.g., epithelioid sarcoma). Treatment naive patients may be enrolled if they have refused standard systemic treatment. Prior adjuvant therapy will not count provided it was completed more than 6 months previously
* Adequate performance status: ECOG 0 or 1/KPS 100-70%
* Adequate organ function determined within 3 weeks of treatment initiation, defined as follows:
* I. Hemoglobin ≥ 8.0 g/dl
* II. Absolute neutrophil count ≥ 1,000/mm^3 (1.0 x 10^9/L)
* III. Platelet count ≥ 75,000/mm3 (75 x 109/L)
* IV. Serum bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for a subject with total bilirubin level > 1.5 x ULN
* V. Aspartate aminotransferase (AST) ≤ 2.5 x ULN OR ≤ 5 x ULN for subjects with liver metastases
* VI. Alanine aminotransferase (ALT) ≤ 2.5 x ULN OR ≤ 5 x ULN for subjects with liver metastases
* VII. Alkaline Phosphatase < 5 x ULN
* VIII. Albumin ≥2.5mg/dL
* IX. Serum creatinine ≤ 1.5 x ULN or a measured or calculateda* creatinine clearance ≥ 60mL/min for subject with creatinine levels > 1.5 x institutional ULN (Note: Creatinine clearance need not be determined if the baseline serum creatinine is within normal limits. GFR can also be used in place of creatinine or CrCl) X. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants XI. Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT and PTT is within therapeutic range of intended use of anticoagulants

  *aCreatinine clearance should be calculated per institutional standard
* Female subject of childbearing potential should have a negative serum pregnancy testing at screening visit and within 72 hours prior to the first dose of study medication

Exclusion Criteria:

* Uncontrolled intercurrent illness including active infection requiring systemic therapy or symptomatic congestive heart failure within 6 months
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrollment. However, in the setting of non-immune mediated indications for use, chronic/active low dose steroid use may be permitted at the discretion of the principal investigator
* Known history of human immunodeficiency virus (HIV) disease
* History or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 years prior to enrollment. Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease
* Active herpetic skin lesions or prior complications of herpetic infection
* Require intermittent or chronic treatment with an intravenous or oral antiherpetic drug (e.g., acyclovir), other than intermittent topical use
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* Received live vaccine or live-attenuated vaccine within 30 days prior to enrollment. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed
* Has a known history of active TB (Bacillus Tuberculosis)
* Female subject is pregnant or breast-feeding, or planning to become pregnant or male subject is planning to father a child within the projected duration of the trial, starting with the pre-screening or screening visit, during study treatment and through 3 months after the last dose of talimogene laherparepvec or 4 months after the last dose of pembrolizumab, whichever is later
* Male and female subjects of childbearing potential who are unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec and 4 months after the last dose of pembrolizumab. (Note: Women not of childbearing potential are defined as: Any female who is post-menopausal [age > 55 years with cessation of menses for 12 or more months or less than 55 years but not spontaneous menses for at least 2 years or less than 55 years and spontaneous menses within the past 1 year, but currently amenorrhoeic(e.g., spontaneous or secondary to hysterectomy), and with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved] or who have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy)
* Sexually active subjects and their partners unwilling to use male or female latex condom or polyurethane condoms for patients with latex allergies to avoid potential viral transmission during sexual contact while on treatment and within 30days after treatment with talimogene laherparepvec
* Subject who is unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or children under the age of 1 year, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec
* Known previous history of sensitivity to talimogene laherparepvec or any of its components to be administered during dosing (e.g. sorbitol, myo-inositol)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Prior therapy with talimogene laherparepvec, tumor vaccine
* Prior chemotherapy, radiotherapy, biological cancer therapy, targeted small molecule therapy or major surgery within 21 days prior to study Day 1 or who has not recovered (i.e., to CTCAE ≤ grade 1 or at baseline) from adverse events due to previously administered therapy. Note: Subjects with ≤ grade 2 neuropathy and alopecia are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Is currently participating and receiving study therapy with another investigational device or study drug or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of the first dose of treatment
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* The presence of any other concurrent active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2026-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ciara Kelly, MBBCh BAO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Enable Medicine (Specimen Analysis Only), Menlo Park, California
  - Stanford University Medical Center, Stanford, California
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center (Data Analysis Only), Houston, Texas

REFERENCES:
- [Derived] Goff PH, Riolobos L, LaFleur BJ, Spraker MB, Seo YD, Smythe KS, Campbell JS, Pierce RH, Zhang Y, He Q, Kim EY, Schaub SK, Kane GM, Mantilla JG, Chen EY, Ricciotti R, Thompson MJ, Cranmer LD, Wagner MJ, Loggers ET, Jones RL, Murphy E, Blumenschein WM, McClanahan TK, Earls J, Flanagan KC, LaFranzo NA, Kim TS, Pollack SM. Neoadjuvant Therapy Induces a Potent Immune Response to Sarcoma, Dominated by Myeloid and B Cells. Clin Cancer Res. 2022 Apr 14;28(8):1701-1711. doi: 10.1158/1078-0432.CCR-21-4239. PMID 35115306
- [Derived] Kelly CM, Antonescu CR, Bowler T, Munhoz R, Chi P, Dickson MA, Gounder MM, Keohan ML, Movva S, Dholakia R, Ahmad H, Biniakewitz M, Condy M, Phelan H, Callahan M, Wong P, Singer S, Ariyan C, Bartlett EK, Crago A, Yoon S, Hwang S, Erinjeri JP, Qin LX, Tap WD, D'Angelo SP. Objective Response Rate Among Patients With Locally Advanced or Metastatic Sarcoma Treated With Talimogene Laherparepvec in Combination With Pembrolizumab: A Phase 2 Clinical Trial. JAMA Oncol. 2020 Mar 1;6(3):402-408. doi: 10.1001/jamaoncol.2019.6152. PMID 31971541
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Talimogene Laherparepvec (T-VEC) Administered With Pembrolizu
Started | 41
Completed | 40
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Talimogene Laherparepvec (T-VEC) Administered With Pembrolizu
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 68 [24 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 28
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Best Objective Response Rate
Description: (complete response + partial response) RECIST 1.1. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Talimogene Laherparepvec (T-VEC) Administered With Pembrolizu
Number analyzed (Participants) | 41
Participants
  Complete Response + Partial Response | 13
  Stable Disease | 13
  Progressive Disease | 14
  Not Evaluable | 1

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Talimogene Laherparepvec (T-VEC) Administered With Pembrolizu
All-Cause Mortality (participants affected / at risk) | 12/41
Serious Adverse Events (participants affected / at risk) | 8/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (T-VEC) Administered With Pembrolizu (N=41)
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, spec (Blood and lymphatic system disorders) | 1
Chills (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 2
Fever (General disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infection (Infections and infestations) | 1
Malaise (General disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Neutrophil count decreased (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Papilledema (Eye disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Uveitis (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (T-VEC) Administered With Pembrolizu (N=41)
Hypoalbuminemia (Metabolism and nutrition disorders) | 33
Hyperglycemia (Metabolism and nutrition disorders) | 31
Anemia (Blood and lymphatic system disorders) | 28
Lymphocyte count decreased (Investigations) | 22
Platelet count decreased (Blood and lymphatic system disorders) | 17
Hypomagnesemia (Metabolism and nutrition disorders) | 16
Alkaline phosphatase increased (Investigations) | 14
Activated partial thromboplastin time prolonged (Investigations) | 13
INR increased (Investigations) | 13
Serum amylase increased (Investigations) | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 12
White blood cell decreased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 11
Hyperkalemia (Metabolism and nutrition disorders) | 10
Lipase increased (Investigations) | 10
Creatinine increased (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 7
Blood bilirubin increased (Investigations) | 5
Neutrophil count decreased (Investigations) | 5
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT03069378/Prot_SAP_000.pdf